CLINICAL TRIAL: NCT05945212
Title: Effects of Local Vibrations Program of Dorsiflexor Muscles on Neuromotor Recovery in Subacute Stroke Patients - a Multicentric Randomized Controlled Study
Brief Title: Effects of Local Vibrations Program of Dorsiflexor Muscles on Neuromotor Recovery in Subacute Stroke Patients.
Acronym: NEUROVIB-AVC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21PH266; 2023-A00489-36 (Other: ANSM)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Stroke Rehabilitation
Keywords: Local vibration; Stroke; Motor recovery; Walking speed; Gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration (Experimental): Stroke patients in subacute rehabilitation phase will be included. In addition of a subacute post-stroke standard rehabilitation program, they will have a vibration program.
  Interventions: Device: Vibration; Other: 10 meters Walk Test; Other: 2 Minute Walk Test (2MWT); Other: Fugl-Meyer (FMA-LE); Other: Modified Ashworth scale; Other: ABILOCO questionnaire; Other: Barthel index; Other: isometric ergometer; Other: Electromyograms (EMG); Other: Traditional quantified gait analysis; Other: SPM - Statistical Parametric Mapping; Other: FACIT questionnaire (Functional Assessment of Chronic Illness Therapy)
- no vibration (Sham Comparator): In addition of a subacute post-stroke standard rehabilitation program, they will have a sham vibration program.
  Interventions: Device: Sham vibration; Other: 10 meters Walk Test; Other: 2 Minute Walk Test (2MWT); Other: Fugl-Meyer (FMA-LE); Other: Modified Ashworth scale; Other: ABILOCO questionnaire; Other: Barthel index; Other: isometric ergometer; Other: Electromyograms (EMG); Other: Traditional quantified gait analysis; Other: SPM - Statistical Parametric Mapping; Other: FACIT questionnaire (Functional Assessment of Chronic Illness Therapy)

INTERVENTIONS:
Device: Vibration — The program will take place over 40 sessions : 5 sessions per week, for 2 months (40 sessions in total over 8 weeks during the hospitalization in the department); this group will benefit from an effective vibration of a frequency of 100Hz
  Other Names: VIBRAMOOV PHYSIO
  Arms: Vibration
Device: Sham vibration — The program will take place over 40 sessions: 5 sessions per week, for 2 months (40 sessions in total over 8 weeks during hospitalization in the department); this group will not benefit from effective vibration.
  Arms: no vibration
Other: 10 meters Walk Test — Short-distance ambulation speed is measurement between 2 markers on the ground 10 meters apart in a corridor with flat ground, the patient starting his walk 3 meters before to have a launched march disregarding markers, and ends 3 meters After. The stopwatch is started when the markers are crossed.
Other: 2 Minute Walk Test (2MWT) — Long-distance ambulation speed is measured from a standing start and the test involves asking the patient to walk as far as possible in 2 minutes.
Other: Fugl-Meyer (FMA-LE) — The Fugl-Meyer (FMA-LE) assessment of motor skills : measurement of the intensity of reflexes, as well as an assessment of voluntary movements and motor coordination. Score from 0 to 34
Other: Modified Ashworth scale — The modified Ashworth scale allows the measurement of spasticity, that is to say the measurement of muscle tone by mobilizing the segment of the lower limb and by evaluating the resistance to stretching of the muscles. Score from 0 to 4
Other: ABILOCO questionnaire — The ABILOCO questionnaire evaluate the autonomy in the walking capacities of the patients (13-items)
Other: Barthel index — The Barthel index measure autonomy in daily life.
Other: isometric ergometer — Evaluate voluntary maximum force in isometric ankle dorsiflexion by Cybex isometric ergometer results.
  Other Names: Cybex isometric ergometer (Henley Healthcare, Sugarland, TX, USA)
Other: Electromyograms (EMG) — Assessment of neuromuscular fatigue by electromyograms (EMG). Surface electrodes is place on the tibial muscle anterior to non-invasively collect electromyograms (EMG). The intensity of stimulation will be gradually increased until a plateau in mechanical (strength) and electromyograms (EMG) responses is obtained.
  Other Names: Electrodes Meditrace 100, Covidien, Mansfield, MA
Other: Traditional quantified gait analysis — Gait kinematics will be recorded on a force platform (90 x 90 cm, Model 9287C, Kistler, Winterthur, Switzerland) to determine: joint angles, net joint moments and powers at the ankle, knee and hip.
  Other Names: 0D
Other: SPM - Statistical Parametric Mapping — Addition of a temporal component to the traditional quantified gait analysis, allowing the focus to be on time series parameters.
  Other Names: 1D
Other: FACIT questionnaire (Functional Assessment of Chronic Illness Therapy) — A short questionnaire consisting of 13 questions to which the patient answers on a scale from 0 to 4. The scores are simply added up, inverting the scale for negative sentences, to give a result out of 52 points. The lower the score, the greater the fatigue.

SUMMARY:
The aim of the vibration intervention proposed in the current study is to allow a better neuromotor recovery in subacute stroke patients when compared with standard rehabilitation alone. These last years, it has been proven that the solicitation of a muscle using vibrations may lead to positive effects on the neuromuscular function. Thus, the aim of the current study is to assess if the addition to a standard rehabilitation program of local vibrations sessions of the dorsiflexor muscles of the paretic limb of stroke patients may allow a better recovery of walking speed (primary outcome). One group using vibrations (i.e. experimental group) and one group with sham vibration (i.e. control group) will take part to this study.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients in subacute rehabilitation phase (between 14 days and 3 months post-stroke)
* Presenting with a stroke, ischemic or hemorrhagic
* Lower-limb deficiency with an initial motor testing < 4 according to the MRC scale
* No neurological history with functional impact other than stroke
* Having received informed information about the study and having signed the written consent
* Affiliated or entitled to a social security scheme.
* Patients under guardianship may be included; they may give their consent with the assistance of their guardian.

If the participant is unable to write, their consent may be given and documented by other appropriate means in the presence of at least one impartial witness. In this case, the witness will sign and date the informed consent document.

Exclusion Criteria:

* Multiple stroke
* Other neurological, cognitive or psychiatric conditions
* Orthopedic ankle history compromising measurements
* Botulinum toxin injected in the lower limb prior the study protocol
* Patient with phlebitis or risk of thrombosis in the lower limb
* Patient under tutorship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Gait speed by 10 meters Walk Test (in meter /second) results | Month 2
  Analysis Gait speed by 10 meters Walk Test (in meter /second) results

SECONDARY OUTCOMES:
Walking performance by 10 meters Walk Test (in meter /second) results | Month 0, 1, 2, 3, 4
  Analysis Walking performance (comfort speed) by 10 meters Walk Test (in meter /second) results
Walking performance by 2 Minute Walk Test (2MWT) (in meter) results | Month 0, 1, 2, 3, 4
  Analysis Walking performance (distance) by 2 Minute Walk Test (2MWT) (in meter) results
Walking performance by Quantified Gait Analysis results | Month 2, 4
  Walking performance will be assessed using: (in m/s) in the 10-meter test (short distance), distance (in m) covered in a 2-minute walk test (long distance) , and qualitatively by a Quantified Gait Analysis (performed only in M2 and M4).
Motor function of the paretic lower limb | Month 4
  The motor function of the paretic lower limb will be measured by the Fugl Meyer Assessment scale for lower limbs (FMA-LE) which includes five domains: Motor skills; Balance skills; Sensitivity; Range of motion; Joint pain. A three-point ordinal scale (0: cannot perform; 1: partially performed; 2: fully performed) is applied to each item. The maximum score is 226.
Lower limb spasticity level | Month 4
  The level of spasticity of the lower limb will be measured by the modified Ashworth scale : a 6-point scale with scores ranging from 0 to 4, where the lowest scores represent normal muscle tone and the highest scores represent spasticity or increased resistance to passive movement.
Autonomy in walking activities | Month 4
  The patient's autonomy in walking activities will be measured by the ABILOCO questionnaire and in daily living activities by the Barthel index.
Lower limb strength | Month 4
  Lower extremity strength will be measured as maximal voluntary strength in isometric ankle dorsiflexion.
Neuromuscular fatigue (1) | Month 4
  Neuromuscular fatigue will be assessed by the level of voluntary activation (in %).
Neuromuscular fatigue (2) | Month 4
  Neuromuscular fatigue will be assessed by corticospinal and intracortical excitability thanks to electromyographic responses evoked by transcranial magnetic stimulation.
Neuromuscular fatigue (3) | Month 4
  Neuromuscular fatigue will be assessed by spinal excitability thanks to electromyographic responses evoked by electrical nerve stimulation.
Neuromuscular fatigue (4) | Month 4
  Neuromuscular fatigue will be assessed by perceived subjective fatigue measured by the FACIT questionnaire : the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System is a collection of health-related quality of life (HRQOL) questionnaires targeted to the management of chronic illness, including over 400 questions. Higher scores for the scales and subscales indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FERNANDEZ, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (7):
- France (7):
  - Centre Hospitalier Georges Claudinon, Le Chambon-Feugerolles
  - Hôpital Marrel, Rive-de-Gier
  - Centre Hospitalier de Roanne, Roanne
  - Service de SSR Val-Rosay, Saint-Didier-au-Mont-d'Or
  - Hôpital Bellevue, CHU de Saint-etienne, Saint-Etienne
  - Service de SSR du Centre Le Clos Champirol, Saint-Etienne
  - Hospices Civils de Lyon, site Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: Yes
Data shared: Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal To achieve aims in the approved proposal Proposals should be directed to corresponding author. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Bessaguet H, Fernandez B, Malejac V, Nerriere E, Velarde M, Coiffet A, Rimaud D, Lapole T. Effect of tibialis anterior focal muscle vibration for gait rehabilitation in hemiplegic individuals during the subacute phase after stroke: the NEUROVIB-AVC study protocol - a multicentric randomised controlled trial. BMJ Open. 2025 May 6;15(5):e102838. doi: 10.1136/bmjopen-2025-102838. PMID 40335131